CLINICAL TRIAL: NCT05241197
Title: Effects of Low-load Resistance Training With Blood Flow Restriction in Patients With Achilles Tendinopathy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Gran Rosario (Other)
Responsible Party: Principal Investigator, Gonzalo Elias, Physiotherapist, University of Gran Rosario
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: BFR and Achilles Tendinopathy
Record Dates: First submitted 2022-02-04; First posted 2022-02-15 (Actual); Last update posted 2024-12-06 (Actual); Status verified 2024-12

CONDITIONS: Achilles Tendinopathy; Achilles Tendon Pain; Tendon Injuries
Keywords: Blood Flow Restriction; Rehabilitation
MeSH Terms: conditions — Tendon Injuries

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Low load training with blood flow restriction (LL-BFR) group. (Experimental): All participants in this arm will use a BFR tourniquet system during the execution of two exercises, unilateral dynamic standing and sitting calf-raises, with a training load of 20% 1 repetition maximum (RM), being progressively increased by 5% every four weeks. Dynamic strength testing will be implemented to re-evaluate the current strength level and adequately adjust the load, using the PowerLift app, which was validated by Balsalobre-Fernandez in 2017. For each exercise, each participant will perform four sets with 30 repetitions the first set and 15 repetitions in the subsequent three sets, counting a total of 75 repetitions. All exercises will be performed in full range of motion (full plantar flexion to full dorsal flexion), with an interset rest period of 1 minute. Three minutes rest was provided between exercises.
  Interventions: Other: Low Load Training with Blood Flow Restriction
- High load training (HLT) group. (Active Comparator): The HLT group will performed the same exercises than the BFR group, however with a training load of 70% 1RM, being progressively increased by 5% every four weeks from 70% to 80%. This protocol will consist of three sets of 6-12 repetitions. Dynamic strength testing will be implemented to re-evaluate the current strength level and adequately adjust the load, using the PowerLift app, which was validated by Balsalobre-Fernandez in 2017. All exercises will be performed in full range of motion, with an interset rest period of 1 minute and a rest period between exercises of 3 minutes.
  Interventions: Other: High Load Training

INTERVENTIONS:
Other: Low Load Training with Blood Flow Restriction — A 12-cm-wide pneumatic nylon tourniquet will be proximally positioned with a snug fit on each thigh. Previously, arterial occlusion pressure (AOP) will be determined using a handheld Doppler Ultrasound in a standing position for each participant. For training routines, cuff pressure will be set to 50% of each individual´s AOP and will be keep inflated during the entire session including the interset rest period of 1 minute. Between the two exercises, the cuff will be deflated for 3 minutes.
  Arms: Low load training with blood flow restriction (LL-BFR) group.
Other: High Load Training — All participants in this arm will do two exercises, unilateral dynamic standing and sitting calf-raises, with a training load of 70% 1RM, being progressively increased by 5% every four weeks from 70% to 80%. This protocol will consist of three sets of 6-12 repetitions with a interset rest period of 1 minute and 3 minutes rest between exercises.
  Arms: High load training (HLT) group.

SUMMARY:
Midportion Achilles tendinopathy (MAT) is a common overuse injury of the lower extremity characterized by the presence of pain, restricted function and interruption of sport activities. Conservative management of MAT has been suggested as the first line of treatment. Actually, there are several exercise programs with beneficial effects on pain and function among which high load training stands out. However, this training modality is inherently difficult to implement in certain populations and pathological conditions due to their inability to tolerate this mechanical stress. In this sense, low load training with blood flow restriction (BFR-LLT) emerges as an effective option in producing hypertrophic adaptations with low intensities (30% 1RM). However, this training modality has not yet been studied in tendon pathology. The aim of this study is to evaluate the potential clinical effects of BFR-LLT in comparison with HLT in patients with chronic MAT.

DETAILED DESCRIPTION:
The aim of this study will be to evaluate the potential clinical effects of low load training with blood flow restriction (BFR-LLT) in comparison with high load training (HLT) in patients with chronic midportion Achilles tendinopathy (MAT). The secondary objectives will be to determine if there are differences in the neovascularity and thickness, pain and function of the AT between both groups in each instance of evaluation. This study will be a simple-blinded randomized clinical trial comprising a total sample size of 52 participants with MAT of both genders and aged between 18 and 50 years. Subjects will undergo a screening process by a sports medicine doctor by different diagnostic tests to identify those presenting a diagnosis of painful MAT and then, they will be randomized into either a group performing HLT (G1), or a group performing BFR-LLT (G2). These volunteers will be recruited in the Parque Hospital (Rosario, Argentine). The study will assess the subjects tendon pain, thickness, cross sectional area and neovascularity, lower limb function, calf raise endurance and jump height. The training protocol will be performed in the University of Gran Rosario (Rosario, Argentine) and will consist of three weekly training sessions during a 12-week rehabilitation period. Primary and secondary outcomes will be measured at baseline, 6 and 12 weeks. All the evaluations will be performed by a blinded physiotherapist.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of unilateral MAT.
* Achilles pain > 3 months.
* Age ranging between 18 to 50 years, both genders.
* Read and speak Spanish well enough to provide informed consent and follow study instructions.
* Can attend in-clinic treatments 2-3 x weekly for the next 12 weeks.

Exclusion Criteria:

* Any ankle or foot surgery.
* History of Achilles rupture.
* Heel pain in the last 3 months.
* Systemic disorders/diseases.
* History of deep venous thrombosis, hypertension or blood clotting disorder.
* Body mass index > 30kg/m2.
* Self-report of pregnancy.
* Drug use (local steroid injection or systemic fluoroquinolones).
* Pain < 2/10 of average pain on NPRS.
* VISA A score > 90%.
* Unable to perform any of the exercises of the study.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 52 (Estimated)
Dates: Start 2022-04-29 (Actual); Primary Completion 2025-11 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Change on pain intensity | At baseline, then at 6 and 12 weeks
  The Numerical Pain Rating Scale (NPRS) will be used to assess pain intensity in daily and sport activities. This scale consists of a sequence of numbers from 0 to 10, in which 0 represents "no pain" and 10 represents "worst pain imaginable".
Change on Victorian Institute of Sport Assessment- Achilles Specific Questionnaire (VISA-A) | At baseline, then at 6 and 12 weeks
  This questionnaire will be used to assess the symptoms, function and pain during daily living and sport activities. The VISA-A consists of 8 questions in which the patients rate the magnitude of pain during rest, function, and activity. The maximum score is 100 points, and a lower score indicates more symptoms and a greater limitation of function and activity.

SECONDARY OUTCOMES:
Change on thickness of the Achilles tendon | At baseline and 12 weeks
  Real time ultrasonography will be performed on the injured Achilles tendon in a longitudinal plane. The thickest point of the tendon will be identified and the A-P distance will be measured (12MHZ linear transducer; Toshiba Aplio300).
Change on cross sectional area of the Achilles tendon | At baseline and 12 weeks
  Real time ultrasonography will be performed on the injured Achilles tendon in a transverse plane. The thickest point of the tendon will be identified and the A-P distance will be measured (12MHZ linear transducer; Toshiba Aplio300).
Change on neovascularization of the Achilles tendon | At baseline and 12 weeks
  Real time ultrasonography with PowerDoppler will be performed in a longitudinal and transverse planes (12MHZ linear transducer; Toshiba Aplio300).
Change on single leg vertical jump | At baseline, then at 6 and 12 weeks
  This test will assess the height in cm, power, strength, velocity and flight time of a vertical jump using the My Jump app, validated by Gallardo-Fuentes in 2016. The instructions will be jumping as high as possible with hands on the subject's waist. Participants will perform 3 repetitions in a non-consecutive manner.
Change on single leg calf-raise endurance test | At baseline, then at 6 and 12 weeks
  This test will assess height, power and work of the calf raise performance during the heel elevation using the Calf Raise app. The test involves going up on the toes and back down as many times the participant can. The test has excellent reliability and is able to detect side-to-side deficits. Participant will be encourage to perform the maximal repetitions during one minute.

CONTACTS AND LOCATIONS:
Overall Officials: Gonzalo Elias, PT, Principal Investigator — University of Gran Rosario
Locations (1):
- University of Gran Rosario, Rosario, Santa Fe Province, Argentina

REFERENCES:
- [Result] Centner C, Lauber B, Seynnes OR, Jerger S, Sohnius T, Gollhofer A, Konig D. Low-load blood flow restriction training induces similar morphological and mechanical Achilles tendon adaptations compared with high-load resistance training. J Appl Physiol (1985). 2019 Dec 1;127(6):1660-1667. doi: 10.1152/japplphysiol.00602.2019. Epub 2019 Nov 14. PMID 31725362
- [Result] Beyer R, Kongsgaard M, Hougs Kjaer B, Ohlenschlaeger T, Kjaer M, Magnusson SP. Heavy Slow Resistance Versus Eccentric Training as Treatment for Achilles Tendinopathy: A Randomized Controlled Trial. Am J Sports Med. 2015 Jul;43(7):1704-11. doi: 10.1177/0363546515584760. Epub 2015 May 27. PMID 26018970
- [Result] Murphy MC, Travers MJ, Chivers P, Debenham JR, Docking SI, Rio EK, Gibson W. Efficacy of heavy eccentric calf training for treating mid-portion Achilles tendinopathy: a systematic review and meta-analysis. Br J Sports Med. 2019 Sep;53(17):1070-1077. doi: 10.1136/bjsports-2018-099934. Epub 2019 Jan 13. PMID 30636702